CLINICAL TRIAL: NCT02556892
Title: Phase 1 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor Ibrutinib in Subjects With Treatment-naive Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Study of Bruton's Tyrosine Kinase (BTK) Inhibitor Ibrutinib in Participants With Treatment-naive Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107620; 54179060LEU1001 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2015-06-30; First posted 2015-09-22 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-07

CONDITIONS: Lymphocytic Leukemia
Keywords: Lymphocytic Leukemia; Ibrutinib; PCI-32765; JNJ-54179060
MeSH Terms: conditions — Leukemia, Lymphoid | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Ibrutinib (Experimental): Participants will self-administer 420 milligram (mg) oral ibrutinib once daily continuously from Cycle 1 to Cycle 6 and thereafter every 28 days until treatment discontinuation.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Participants will self-administer 420 milligram (mg) oral ibrutinib once daily continuously from Cycle 1 to Cycle 6 and thereafter every 28 days until treatment discontinuation.
  Other Names: PCI-32765; JNJ-54179060

SUMMARY:
The purpose of this study is to evaluate the safety of Ibrutinib in Japanese participants with treatment-naive chronic lymphocytic leukemia ( CLL) or small lymphocytic lymphoma (SLL).

DETAILED DESCRIPTION:
This is a Phase 1, open-label and multicenter study. The study consists of a Screening Phase (28 days prior to the first administration of the study drug), Treatment Phase (time when the first dose of ibrutinib is administered until disease progression, the investigator no longer considers the treatment to be tolerable, or the participant meets any one of the discontinuation criteria) and Follow-up Phase (end of the last dose of study drug until 30 days after the last dose of study drug or the start of subsequent anti-CLL/SLL therapy, whichever comes first). Participants will be instructed to take 3 capsules of ibrutinib (at a dose of 420 mg) orally once daily starting at Cycle 1, Day 1. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that meets published diagnostic criteria
* For CLL participants: Measurable nodal disease by computed tomography (CT), defined as at least 1 lymph node greater than (>) 1.5 centimeter (cm) at the longest diameter at a site that has not been previously irradiated. Adequate hepatic function, defined as serum aspartate transaminase (AST) and alanine; For SLL participants: At least 1 measurable site of disease according to the Revised Response Criteria for Malignant Lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate hepatic function, defined as serum aspartate transaminase (AST) and alanine transaminase (ALT) <2.5 × upper limit of normal (ULN), and total bilirubin less than or equal to (<=) 1.5 × ULN (unless due to Gilbert's syndrome)
* A woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening

Exclusion Criteria:

* Known involvement of the central nervous system by lymphoma or leukemia
* History or current evidence of Richter's transformation or prolymphocytic leukemia
* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura
* Any previous treatment (chemotherapy, radiotherapy, and/or monoclonal antibodies) intended specifically to treat CLL/SLL
* Received any immunotherapy, live vaccine, or investigational drug within 4 weeks prior to the first dose of the study drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07-03 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Intensity of Adverse Events (AEs) | Screening up to follow-up phase (maximum of 24 months)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Intensity of Adverse Events will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).
Incidence of Adverse Events | Screening up to follow-up phase (maximum of 24 months)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Incidence was defined as the number of participants who experienced an adverse event within their period of participation in this study. Incidence of adverse events will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE).

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve (AUC) Over the Dosing Interval | Pre-dose and 1, 2, and 4 hours post-dose on Day 1 of Cycle 1 and Cycle 2
Overall Response Rate (Complete Response [CR] and Partial Response [PR]) | Days 1 of cycles 3,5,7 and every odd numbered cycle thereafter until disease progression, unacceptable toxicity or death whichever is first; expected average of 24 months
  Tumor response will be evaluated according to the Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia (CLL) and the International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma, respectively.
Time to Response | Days 1 of cycles 3,5,7 and every odd numbered cycle thereafter until disease progression, unacceptable toxicity or death whichever is first; expected average of 24 months
  Time to response is defined as the time from the initial treatment until the first documented evidence of CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (8):
- Japan (8):
  - Fukuoka
  - Hiroshima
  - Isehara
  - Kobe
  - Kōtoku
  - Osaka
  - Sapporo
  - Tachikawa

REFERENCES:
- See also: Phase 1 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor Ibrutinib in Subjects With Treatment-naive Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR107620&attachmentIdentifier=2d0a9e6d-8e4a-4ec2-a334-bf738f197d66&fileName=CR107620_CSR_Synopsis.pdf&versionIdentifier=